CLINICAL TRIAL: NCT03766399
Title: A Single-blind, Randomized, Placebo-Controlled 3-Part Study in Healthy Volunteers and Patients With Mild Asthma to Investigate the Safety, Tolerability and Pharmacokinetics of Inhaled AZD0449 Following Single and Multiple Ascending Doses and to Investigate the Anti-Inflammatory Effect of Inhaled AZD0449
Brief Title: A Study in Healthy Volunteers and Patients With Mild Asthma to Investigate the Safety, Anti-inflammatory Effect of Inhaled AZD0449
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: D5371C00001; 2018-003469-32 (EudraCT Number)
Record Dates: First submitted 2018-11-08; First posted 2018-12-06 (Actual); Results first posted 2024-08-23 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-03

CONDITIONS: Asthma
Keywords: Inhaled JAK inhibitor
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (13):
- Part 1a (SAD) Cohort 1 (Experimental): 6 participants will receive inhaled dose 1 of AZD0449 nebulized suspension and 2 participants will receive inhaled placebo.
  Interventions: Drug: AZD0449; Drug: Placebo
- Part 1a (SAD) Cohort 2 (Experimental): 6 participants will receive inhaled dose 2 of AZD0449 nebulized suspension and 2 participants will receive inhaled placebo.
  Interventions: Drug: AZD0449; Drug: Placebo
- Part 1a (SAD) Cohort 3 (Experimental): 6 participants will receive inhaled dose 3 of AZD0449 nebulized suspension and 2 participants will receive inhaled placebo.
  Interventions: Drug: AZD0449; Drug: Placebo
- Part 1a (SAD) Cohort 4 (Experimental): 6 participants will receive inhaled dose 4 of AZD0449 nebulized suspension and 2 participants will receive inhaled placebo.
  Interventions: Drug: AZD0449; Drug: Placebo
- Part 1a (SAD) Cohort 5 (Placebo Comparator): 6 participants will receive inhaled dose 5 of AZD0449 nebulized suspension and 2 participants will receive inhaled placebo.
  Interventions: Drug: AZD0449; Drug: Placebo
- Part 1a (SAD) Cohort 6 (Experimental): 6 participants will receive inhaled dose 6 of AZD0449 nebulized suspension and 2 participants will receive inhaled placebo.
  Interventions: Drug: AZD0449; Drug: Placebo
- Part 1b (IV cohort 1) (Experimental): All 6 participants will receive single IV dose of AZD0449 solution.
  Interventions: Drug: AZD0449; Drug: Placebo
- Part 2a (MAD) Cohort 1 (Experimental): 6 participants will receive inhaled dose 7 of AZD0449 nebulized suspension and 3 participants will receive inhaled placebo.
  Interventions: Drug: AZD0449; Drug: Placebo
- Part 2a (MAD) Cohort 2 (Experimental): 6 participants will receive inhaled dose 8 of AZD0449 nebulized suspension and 3 participants will receive inhaled placebo.
  Interventions: Drug: AZD0449; Drug: Placebo
- Part 2b (MAD/healthy volunteers) Cohort 3 (Experimental): 18 healthy volunteers will receive inhaled dose 9 of AZD0449 nebulized suspension and 12 healthy volunteers will receive inhaled placebo.
  Interventions: Drug: AZD0449; Drug: Placebo
- Part 3a (DPI/PoM) (Experimental): 18 participants will receive inhaled dose 10 of AZD0449 DPI and 6 participants will receive inhaled placebo.
  Interventions: Drug: AZD0449; Drug: Placebo
- Part 1b (IV cohort 2) (Experimental): 6 healthy volunteers will receive single IV dose of AZD0449 solution.
  Interventions: Drug: AZD0449; Drug: Placebo
- Part 3b (DPI/healthy volunteers) (Experimental): Part 3b is optional. 8 healthy volunteers; 6 volunteers will receive AZD0449 DPI and 2 volunteers will recieve placebo.
  Interventions: Drug: AZD0449; Drug: Placebo

INTERVENTIONS:
Drug: AZD0449 — Participants will receive single inhaled AZD0449 nebulizer suspension and single IV dose of AZD0449 solution.
Drug: Placebo — Participants will receive single dose of placebo for AZD0449 (nebulizer suspension).

SUMMARY:
This will be a Phase I, first in human (FIH) study consisting of the following parts: Part 1a (SAD), Part 1b (IV Cohort), Part 2 (Multiple ascending dose (MAD), and Part 3 dry-powder inhalation (DPI)/ Proof of mechanism (PoM). Part 1a of the study will be a randomized, single-blind, placebo-controlled, SAD, sequential group design study performed at a single study center. Part 1b, will be an open-label, single-dose, single-cohort study. It will follow a 2-stage design in the way that participants from Part 1a will be selected for the IV Cohort in Part 1b. Part 2 of the study will be a randomized, single-blind, placebo-controlled, MAD, sequential group design and study performed at 3 study centers. Part 3a/b will be a randomized, single-blind, placebo-controlled, DPI/PoM study. The expected duration of each subject in Part 1a of the study is up to 36 days and up to 53 days for subjects participating in Part 1b. The expected duration of each participant in Part 2 is up to 52 days and Part 3 is up to 55 days.

DETAILED DESCRIPTION:
This will be a Phase I, consisting of the following parts: Part 1a, Part 1b, Part 2a/b, Part 3a/b. Part 1a of the study will be a randomized, single-blind, placebo-controlled, SAD, sequential group design study performed at a single study center. Six inhaled dose levels of AZD0449 nebulized suspension are planned to be investigated in 6 cohorts. Depending on emerging safety and PK data, up to 3 additional inhaled dose levels (cohorts), within the pre-specified dose range, may be added at the discretion of the Sponsor. Within each cohort, 6 volunteers will be randomized to receive an inhaled dose of AZD0449 nebulized suspension and 2 volunteers will be randomized to receive inhaled placebo. Intravenous (IV) dosing in Part 1b of the study will be initiated after the completion of cohort 6 in Part 1a or (if Part 1a is completed with less than 6 cohorts) after completion of the last cohort in Part 1a. Part 1b, will be open-label and consist of 2 dose cohorts (IV 0.090 mg and 0.360 mg) and be conducted in 12 healthy volunteers. Six (6) volunteers will be selected for the first IV dose cohort in Part 1b following a 2-stage design. If Part 1b cannot be completed with 6 volunteers from Part 1a or if some of the data are considered not evaluable, up to 6 additional naïve volunteers may be enrolled. A second IV dose cohort in Part 1b will be initiated after the evaluation of the PK and safety results from all cohorts in Part 1a and completion of the first IV dose cohort in Part 1b. The second IV dose cohort will consist of 6 healthy volunteers who have not previously participated in the study (naïve volunteers). Part 2a/b of the study will be a randomized, single-blind, placebo-controlled, MAD, sequential group design study performed at approximately 3 study centers. Part 2a will include cohorts 1 and 2, each comprising of 9 patients with mild asthma. Within each of these cohorts 6 patients will be randomized to receive AZD0449 nebulized suspension and 3 patients randomized to receive placebo. Additional cohorts with 9 patients could be added to study PK, PD and safety for doses lower than 1.2 mg or up to 5 mg. Part 2b will consist of 1 cohort of 8 healthy volunteers; 6 volunteers will be randomized to receive AZD0449 nebulized suspension and 2 volunteers will be randomized to receive placebo. Part 3a/b of the study will be initiated after the completion of Part 2b. Part 3a/b will be a randomized, single-blind, placebo-controlled, DPI/PoM study. Part 3 will be conducted in up to 36 patients with mild asthma (Part 3a) and 8 healthy volunteers (Part 3b, optional). Part 3a will consist of 36 patients, where 18 patients will be randomized to AZD0449 DPI and 18 patients to placebo. An Interim Analysis (IA) will be conducted when 9 patients on each arm have completed the study (50% Part 3a). Should new data on the variability of the FeNO measurements emerge at the IA, the sample size in Part 3a could be changed. If the optional Part 3b is conducted, it will comprise 8 healthy volunteers; 6 volunteers will be randomized to AZD0449 DPI and 2 volunteers to placebo.

ELIGIBILITY:
Inclusion criteria:

Part 1a/b: 1. Provision of signed and dated, written informed consent before any study specific procedures (applicable for all parts). 2. Healthy male volunteers and healthy female volunteers (for Part 1a and Part 1b first IV cohort, female volunteers must be of non-childbearing potential), aged 18 to 55 years with suitable veins for cannulation or repeated venipuncture. 3. Female patients must not be lactating and must have a negative pregnancy test at the Screening Visit and on admission to the Clinical Unit. Women of non-childbearing potential must fulfill one of the following criteria (Applicable for all parts): 3.1. Postmenopausal defined as amenorrhea for at least 12 months or more following cessation of all exogenous hormonal treatments and follicle-stimulating hormone (FSH) levels in the postmenopausal range. 3.2. Documentation of irreversible surgical sterilization by hysterectomy, bilateral oophorectomy or bilateral salpingectomy but not tubal ligation. 4. Have a body mass index (BMI) between 18 and 30 kg/m2 inclusive and weigh at least 60 kg. 5. Healthy volunteer has a Forced Expiratory Volume in one second (FEV1) ≥80% of the predicted value regarding age, height, gender and ethnicity at the Screening Visit. 6. Male volunteers and their WOCBP partners should be willing to use highly effective contraception measures and should refrain from donating sperm or fathering a child from the first day of dosing until 3 months after the last dose of IMP. 7. Female volunteers in Part 1b second IV cohort should be willing to use highly effective contraception measures from the first day of dosing until 1 month after the last dose of IMP. 8. Provision of signed, written and dated informed consent for optional genetic research. If a volunteer declines to participate in the genetic component of the study, there will be no penalty or loss of benefit to the volunteer. The volunteer will not be excluded from other aspects of the study described in this protocol. Patients with mild asthma (Part 2a and Part 3a): 1. Male and female (including WOCBP) patients with mild asthma aged 18 to 55 years with suitable veins for cannulation or repeated venipuncture. 2. Patients must be willing to remain in house at the study center for 16 consecutive days (part 2a) or for 30 consecutive days, optional from Day 17 for Germany (part 3a). 3. Have a BMI between 18 and 35 kg/m2 inclusive and weigh at least 50 kg. 4. Physician diagnosed (mild) asthma for at least 6 months prior to screening. 5. Lung function ≥70% predicted for Forced Expiratory Volume in 1 second (FEV1) at the Screening Visit AND at the 12 h timepoint on Day -1, in accordance with the American Thoracic Society (ATS)/European Respiratory Society (ERS) criteria. 6. Have a FeNO of ≥30 ppb at the Screening Visit and at the 12 h timepoint on Day -1. 7. Male patients and their WOCBP partners should be willing to use highly effective contraception measures and should refrain from donating sperm or fathering a child from the first day of dosing until 3 months after the last dose of IMP (applicable for part 2b and 3b). 8. Female patients should be willing to use highly effective contraception measures from the first day of dosing until 1 month after the last dose of IMP. 9. Provision of signed, written and dated informed consent for optional genetic research. If a patient declines to participate in the genetic component of the study, there will be no penalty or loss of benefit to the patient. The patient will not be excluded from other aspects of the study described in this protocol.

Healthy volunteers (Part 2b and Part 3b): 1. Healthy male and female (including WOCBP) volunteers aged 18 to 55 years with suitable veins for cannulation or repeated venipuncture. 2. Have a BMI between 18 and 30 kg/m2 inclusive and weigh at least 60 kg. 3. Healthy volunteer has a Forced Expiratory Volume in one second (FEV1) ≥80% of the predicted value regarding age, height, gender and ethnicity at the Screening Visit and at the 12 h timepoint on Day -1, in accordance with the ATS/ERS criteria. 4. Female volunteers should be willing to use highly effective contraception measures from the first day of dosing until 1 month after the last dose of IMP. 5. Provision of signed, written and dated informed consent for optional genetic research. If a healthy volunteer declines to participate in the genetic component of the study, there will be no penalty or loss of benefit to the healthy volunteer. The healthy volunteer will not be excluded from other aspects of the study described in this protocol.

Exclusion criteria:

Part 1a/b: 1. History of any clinically important disease or disorder which, in the opinion of the Investigator, may either put the volunteer at risk because of participation in the study, or influence the results or the volunteer's ability to participate in the study. 2. History of any respiratory disorders such as asthma, chronic obstructive pulmonary disease (COPD) or idiopathic pulmonary fibrosis (IPF) (applicable for all parts). 3. Healthy volunteer has an increased risk of infection. 4. History or presence of gastrointestinal, hepatic or renal disease or any other condition known to interfere with absorption, distribution, metabolism or excretion of drugs (applicable to all parts). 5. Any clinically important illness, medical/surgical procedure or trauma within 4 weeks of the first administration of IMP (applicable to all parts). 6. Any laboratory values with the following deviations at the Screening Visit and on admission to the Clinical Unit. Abnormal values may be repeated once at the discretion of the Investigator (applicable to all parts): 6.1. Alanine aminotransferase (ALT) >upper limit of normal (ULN). 6.2. Aspartate aminotransferase (AST) >ULN. 6.3. Creatinine >ULN. 6.4. White blood cell (WBC) count <LLN (Lower limit of normal). 6.5. Hemoglobin <LLN. 7. Any clinically important abnormalities in clinical chemistry, hematology or urinalysis results, other than those described under exclusion criteria numbers 3 and 6, as judged by the Investigator (Applicable to all parts). 8. Abnormal vital signs, after 10 minutes supine rest. Abnormal values may be repeated once at the discretion of the Investigator (applicable to all parts). 9. Any clinically important abnormalities in rhythm, conduction or morphology of the resting ECG and any clinically important abnormalities in the 12-lead electrocardiogram (ECG) as considered by the Investigator that may interfere with the interpretation of QTc interval changes, including abnormal ST-T-wave morphology, particularly in the protocol defined primary lead or left ventricular hypertrophy at the Screening Visit and Day -1 (Applicable to all parts). 10. Known or suspected history of drug abuse [within the past 2 years for Part 2a and Part 3a] as judged by the Investigator (Applicable to all parts). 11.Current smokers or those who have smoked or used nicotine products (including e-cigarettes) within the previous 6 months or has smoking history of >5 pack-years (applicable to all parts). 12. History of alcohol abuse or excessive intake of alcohol as judged by the Investigator (in Germany only: excessive intake of alcohol defined as the regular consumption of more than 3 units [24 g] of alcohol per day for men or 2 units [16 g] of alcohol per day for women) (Applicable to all parts). 13. Positive screen for drugs of abuse, cotinine (nicotine) or alcohol at the Screening Visit or on admission to the Clinical Unit (Applicable to all parts). 14. History of severe allergy/hypersensitivity or ongoing clinically important allergy/hypersensitivity, as judged by the Investigator or history of hypersensitivity to drugs with a similar chemical structure or class to AZD0449 (Applicable to all parts). 15. Use of drugs with enzyme inducing properties such as St John's Wort within 3 weeks before the first administration of IMP (Applicable to all parts). 16. Plasma donation within 1 month of the Screening Visit or any blood donation/blood loss >500 mL during the 3 months before the Screening Visit (Applicable to all parts). 17. Healthy volunteers/patients who have previously received (Applicable to all parts). 18. Involvement of any AstraZeneca or Clinical Unit employee or their close relatives (Applicable to all parts). Patients with mild asthma (Part 2a and Part 3a): 1. History of any clinically important disease other than asthma, or disorder which, in the opinion of the Investigator, may either put the patient at risk because of participation in the study, or influence the results or the patient's ability to participate in the study. 2. Patient has an increased risk of infection. 3. Suspicion of Gilbert's syndrome. 4. Exacerbation of asthma symptoms within 6 months prior to Screening and Day -1 and requiring the use of oral or IV steroids, antibiotics, Accident and Emergency visit, or hospital admission to the Clinical Unit. 5. Female patients who are pregnant, breastfeeding, or are planning a pregnancy during the study period or within 1 month after the last dose of IMP. Healthy volunteers (Part 2b and Part 3b): 1.History of any clinically important disease or disorder which, in the opinion of the Investigator, may either put the volunteer at risk because of participation in the study, or influence the results or the volunteer's ability to participate in the study. 2. Female healthy volunteers who are pregnant, breastfeeding, or are planning a pregnancy during the study period or within 1 month after the last dose of IMP.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2018-11-30 (Actual); Primary Completion 2021-06-24 (Actual); Study Completion 2021-06-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dave Singh, Principal Investigator — The Medicines Evaluation Unit
Locations (4):
- Research Site, Berlin, Germany
- Research Site, Wellington, New Zealand
- United Kingdom (2):
  - Research Site, Harrow
  - Research Site, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5371C00001&attachmentIdentifier=f7a8a707-e4fc-4d6d-bed0-6383d9f8cae5&fileName=AZ_D5371c00001_(PXL_240729)__CSR_Synopsis_Final_Draft_to_Client_Redacted.pdf&versionIdentifier=
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5371C00001&attachmentIdentifier=1c10d56d-06fb-4ddb-9518-f952f8030717&fileName=AZ_D5371c00001_(PXL_240729)__Protocol_Final_Draft_to_Client_Redacted.pdf&versionIdentifier=
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5371C00001&attachmentIdentifier=e3227c6b-8a65-42e9-9a1d-9d5b7464ae3f&fileName=AZ_D5371c00001_(PXL_240729)__SAP_Final_Draft_to_Client_Redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was a 3 part study conducted between 30 Nov 2018 and 24 Jun 2021. Part 1 was conducted at a single clinical unit. Part 2 was conducted at 3 clinical units.
Pre-assignment Details: Part 1a was a single ascending dose (SAD) study in healthy participants. Part 1b consisted of 2 IV dose cohorts. 6 participants from Part 1a in first IV dose cohort and 6 healthy participants in second IV dose cohort were selected for Part 1b. Part 2 was a multiple ascending dose (MAD) study in patients with mild asthma (Part 2a) and healthy participants (Part 2b). Part 3 included patients with mild asthma (Part 3a) and healthy participants (Part 3b).
Groups:
- Part 1a (SAD) Placebo; Part 2b (MAD) Placebo; Part 3b (DPI/Healthy Participants) Placebo: Randomized healthy participants received Placebo for AZD0449.
- Part 1a (SAD) Cohort 1: Randomized healthy participants received a single inhaled dose of AZD0449 0.095 mg nebulized suspension via Jet nebulizer.
- Part 1a (SAD) Cohort 2: Randomized healthy participants received a single inhaled dose of AZD0449 0.28 mg nebulized suspension via Jet nebulizer.
- Part 1a (SAD) Cohort 3: Randomized healthy participants received a single inhaled dose of AZD0449 0.84 mg nebulized suspension via Jet nebulizer.
- Part 1a (SAD) Cohort 4: Randomized healthy participants received a single inhaled dose of AZD0449 1.60 mg nebulized suspension via Jet nebulizer.
- Part 1a (SAD) Cohort 5: Randomized healthy participants received a single inhaled dose of AZD0449 3.20 mg nebulized suspension via Jet nebulizer.
- Part 1a (SAD) Cohort 6: Randomized healthy participants received a single inhaled dose of AZD0449 5 mg nebulized suspension via Jet nebulizer.
- Part 1b (SAD IV) Cohort 1: Randomized healthy participants received a single intravenous (IV) dose of AZD0449 0.090 mg solution.
- Part 1b (SAD IV) Cohort 2: Randomized healthy participants received a single IV dose of AZD0449 0.360 mg solution.
- Part 2a (MAD) Placebo: Randomized patients with mild asthma received Placebo.
- Part 2a (MAD) Cohort 1: Randomized patients with mild asthma received a multiple inhaled dose of AZD0449 1.20 mg nebulized suspension via Jet nebulizer.
- Part 2a (MAD) Cohort 2: Randomized patients with mild asthma received a multiple inhaled dose of AZD0449 2.50 mg nebulized suspension via Jet nebulizer.
- Part 2b (MAD) Cohort 1: Randomized healthy participants received a multiple inhaled of AZD0449 5 mg nebulized suspension via Jet nebulizer.
- Part 3a (DPI/PoM) Placebo: Randomized patients with mild asthma received Placebo for AZD0449.
- Part 3a Dry Powder Inhalation/Proof of Mechanism (DPI/PoM): Randomized patients with mild asthma received a multiple inhaled dose of AZD0449 5 mg DPI.
- Part 3b (DPI/Healthy Participants): Randomized healthy participants received multiple inhaled dose of AZD0449 5 mg DPI.
Period: Part 1a: SAD (Nebulized Inhalation)
Arm/Group | Part 1a (SAD) Placebo | Part 1a (SAD) Cohort 1 | Part 1a (SAD) Cohort 2 | Part 1a (SAD) Cohort 3 | Part 1a (SAD) Cohort 4 | Part 1a (SAD) Cohort 5 | Part 1a (SAD) Cohort 6 | Part 1b (SAD IV) Cohort 1 | Part 1b (SAD IV) Cohort 2 | Part 2a (MAD) Placebo | Part 2a (MAD) Cohort 1 | Part 2a (MAD) Cohort 2 | Part 2b (MAD) Placebo | Part 2b (MAD) Cohort 1 | Part 3a (DPI/PoM) Placebo | Part 3a Dry Powder Inhalation/Proof of Mechanism (DPI/PoM) | Part 3b (DPI/Healthy Participants) Placebo | Part 3b (DPI/Healthy Participants)
Started | 12 | 6 | 6 | 6 | 6 | 6 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 12 | 6 | 6 | 6 | 6 | 6 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 1b: SAD (Intravenous Dosing)
Arm/Group | Part 1a (SAD) Placebo | Part 1a (SAD) Cohort 1 | Part 1a (SAD) Cohort 2 | Part 1a (SAD) Cohort 3 | Part 1a (SAD) Cohort 4 | Part 1a (SAD) Cohort 5 | Part 1a (SAD) Cohort 6 | Part 1b (SAD IV) Cohort 1 | Part 1b (SAD IV) Cohort 2 | Part 2a (MAD) Placebo | Part 2a (MAD) Cohort 1 | Part 2a (MAD) Cohort 2 | Part 2b (MAD) Placebo | Part 2b (MAD) Cohort 1 | Part 3a (DPI/PoM) Placebo | Part 3a Dry Powder Inhalation/Proof of Mechanism (DPI/PoM) | Part 3b (DPI/Healthy Participants) Placebo | Part 3b (DPI/Healthy Participants)
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 2a: MAD (Nebulized Inhalation)
Arm/Group | Part 1a (SAD) Placebo | Part 1a (SAD) Cohort 1 | Part 1a (SAD) Cohort 2 | Part 1a (SAD) Cohort 3 | Part 1a (SAD) Cohort 4 | Part 1a (SAD) Cohort 5 | Part 1a (SAD) Cohort 6 | Part 1b (SAD IV) Cohort 1 | Part 1b (SAD IV) Cohort 2 | Part 2a (MAD) Placebo | Part 2a (MAD) Cohort 1 | Part 2a (MAD) Cohort 2 | Part 2b (MAD) Placebo | Part 2b (MAD) Cohort 1 | Part 3a (DPI/PoM) Placebo | Part 3a Dry Powder Inhalation/Proof of Mechanism (DPI/PoM) | Part 3b (DPI/Healthy Participants) Placebo | Part 3b (DPI/Healthy Participants)
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6 | 6 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6 | 6 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 2b: MAD (Nebulized Inhalation)
Arm/Group | Part 1a (SAD) Placebo | Part 1a (SAD) Cohort 1 | Part 1a (SAD) Cohort 2 | Part 1a (SAD) Cohort 3 | Part 1a (SAD) Cohort 4 | Part 1a (SAD) Cohort 5 | Part 1a (SAD) Cohort 6 | Part 1b (SAD IV) Cohort 1 | Part 1b (SAD IV) Cohort 2 | Part 2a (MAD) Placebo | Part 2a (MAD) Cohort 1 | Part 2a (MAD) Cohort 2 | Part 2b (MAD) Placebo | Part 2b (MAD) Cohort 1 | Part 3a (DPI/PoM) Placebo | Part 3a Dry Powder Inhalation/Proof of Mechanism (DPI/PoM) | Part 3b (DPI/Healthy Participants) Placebo | Part 3b (DPI/Healthy Participants)
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 7 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 6 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Period: Part 3a: Asthma Patients (DPI)
Arm/Group | Part 1a (SAD) Placebo | Part 1a (SAD) Cohort 1 | Part 1a (SAD) Cohort 2 | Part 1a (SAD) Cohort 3 | Part 1a (SAD) Cohort 4 | Part 1a (SAD) Cohort 5 | Part 1a (SAD) Cohort 6 | Part 1b (SAD IV) Cohort 1 | Part 1b (SAD IV) Cohort 2 | Part 2a (MAD) Placebo | Part 2a (MAD) Cohort 1 | Part 2a (MAD) Cohort 2 | Part 2b (MAD) Placebo | Part 2b (MAD) Cohort 1 | Part 3a (DPI/PoM) Placebo | Part 3a Dry Powder Inhalation/Proof of Mechanism (DPI/PoM) | Part 3b (DPI/Healthy Participants) Placebo | Part 3b (DPI/Healthy Participants)
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 18 | 18 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 18 | 18 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 3b: Healthy Participants (DPI)
Arm/Group | Part 1a (SAD) Placebo | Part 1a (SAD) Cohort 1 | Part 1a (SAD) Cohort 2 | Part 1a (SAD) Cohort 3 | Part 1a (SAD) Cohort 4 | Part 1a (SAD) Cohort 5 | Part 1a (SAD) Cohort 6 | Part 1b (SAD IV) Cohort 1 | Part 1b (SAD IV) Cohort 2 | Part 2a (MAD) Placebo | Part 2a (MAD) Cohort 1 | Part 2a (MAD) Cohort 2 | Part 2b (MAD) Placebo | Part 2b (MAD) Cohort 1 | Part 3a (DPI/PoM) Placebo | Part 3a Dry Powder Inhalation/Proof of Mechanism (DPI/PoM) | Part 3b (DPI/Healthy Participants) Placebo | Part 3b (DPI/Healthy Participants)
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 6
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Part 3a (DPI/PoM): Randomized patients with mild asthma received a multiple inhaled dose of AZD0449 5 mg DPI.
- Total: Total of all reporting groups
Arm/Group | Part 1a (SAD) Placebo | Part 1a (SAD) Cohort 1 | Part 1a (SAD) Cohort 2 | Part 1a (SAD) Cohort 3 | Part 1a (SAD) Cohort 4 | Part 1a (SAD) Cohort 5 | Part 1a (SAD) Cohort 6 | Part 1b (SAD IV) Cohort 1 | Part 1b (SAD IV) Cohort 2 | Part 2a (MAD) Placebo | Part 2a (MAD) Cohort 1 | Part 2a (MAD) Cohort 2 | Part 2b (MAD) Cohort 1 | Part 2b (MAD) Placebo | Part 3a (DPI/PoM) | Part 3a (DPI/PoM) Placebo | Part 3b (DPI/Healthy Participants) Placebo | Part 3b (DPI/Healthy Participants) | Total
Number analyzed (Participants) | 12 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 7 | 2 | 18 | 18 | 2 | 6 | 131
Age, Continuous [Mean (Standard Deviation); unit: Years] | 31.7 (8.1) | 29.8 (6.6) | 29.3 (7.6) | 36.3 (7.7) | 26.3 (5.5) | 35.8 (10.1) | 30.7 (10.4) | 32.8 (7.5) | 28.5 (4.0) | 37.5 (8.5) | 35.7 (13.7) | 38.7 (13.5) | 41.1 (9.4) | 33.0 (11.3) | 30.0 (9.2) | 30.2 (9.1) | 48.0 (4.2) | 36.8 (14.5) | 32.8 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 2 | 0 | 0 | 9 | 8 | 0 | 2 | 25
  Male | 12 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 2 | 6 | 6 | 4 | 7 | 2 | 9 | 10 | 2 | 4 | 106
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 5
  Not Hispanic or Latino | 12 | 6 | 6 | 4 | 6 | 6 | 6 | 6 | 6 | 5 | 6 | 6 | 7 | 2 | 18 | 16 | 2 | 6 | 126
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 10 | 4 | 2 | 4 | 4 | 5 | 4 | 3 | 5 | 4 | 5 | 5 | 7 | 1 | 13 | 14 | 2 | 5 | 97
  Black or African American | 0 | 1 | 3 | 1 | 1 | 1 | 1 | 3 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 14
  Asian | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 1 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  American Indian or Alaska native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Other | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 2 | 0 | 0 | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events and Serious Adverse Events
Description: Safety and tolerability of AZD0449 following inhaled administration of single ascending doses to healthy participants, inhaled nebulized administration of multiple ascending doses to healthy participants and patients with mild asthma, and repeated inhaled administration to patients with mild asthma using a DPI was assessed.
Time Frame: From screening up to follow-up visit [Part 1 a (6±1 Days post-dose)] [Part 2a (Day 22±1 (10±1 days post-last dose)], Safety Monitoring Period 2b/3a [Day 17 to 27 (15 day post-last dose)]
Population: Safety Analysis Set included all participants and patients who received at least one dose of AZD0449 and for whom any safety post-dose data were available.
Measure: Number; unit: Participants
Arm/Group | Part 1a (SAD) Placebo | Part 1a (SAD) Cohort 1 | Part 1a (SAD) Cohort 2 | Part 1a (SAD) Cohort 3 | Part 1a (SAD) Cohort 4 | Part 1a (SAD) Cohort 5 | Part 1a (SAD) Cohort 6 | Part 2a (MAD) Placebo | Part 2a (MAD) Cohort 1 | Part 2a (MAD) Cohort 2 | Part 2b (MAD) Placebo | Part 2b (MAD) Cohort 1 | Part 3a (DPI/PoM) Placebo | Part 3a (DPI/PoM) | Part 3b (DPI/Healthy Participants) Placebo | Part 3b (DPI/Healthy Participants)
Number analyzed (Participants) | 12 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 2 | 7 | 18 | 18 | 2 | 6
Participants
  Any Adverse Event (AE) | 3 | 2 | 2 | 3 | 3 | 3 | 1 | 4 | 5 | 3 | 2 | 6 | 15 | 14 | 0 | 3
  Any AE with outcome=death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any serious AE (including events with outcome=death) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any AE leading to withdrawal from study | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Any AE leading to discontinuation of investigational medicinal product (IMP) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

2. Primary Outcome: Maximum Observed Plasma Concentration (Cmax)
Description: Cmax of AZD0449 following intravenous administration of a single dose to healthy participants was assessed.
Time Frame: Part 1b: Day 1
Population: The pharmacokinetic (PK) set consisted of all participants who received at least one dose of AZD0449 and who had evaluable PK data, with no major protocol deviations thought to impact on the analysis of the PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomole/liter (nmol/L)
Arm/Group | Part 1b (SAD IV) Cohort 1 | Part 1b (SAD IV) Cohort 2
Number analyzed (Participants) | 6 | 6
nanomole/liter (nmol/L) | 2.053 (15.95) | 10.31 (17.58)

3. Primary Outcome: Area Under the Plasma Concentration Time Curve From Time Zero to Infinity (AUCinf)
Description: AUCinf of AZD0449 following intravenous administration of a single dose to healthy participants was assessed.
Time Frame: Part 1b: Day 1
Population: The PK set consisted of all participants who received at least one dose of AZD0449 and who had evaluable PK data, with no major protocol deviations thought to impact on the analysis of the PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*nmol/L
Arm/Group | Part 1b (SAD IV) Cohort 1 | Part 1b (SAD IV) Cohort 2
Number analyzed (Participants) | 6 | 6
h*nmol/L | 3.697 (14.27) | 17.10 (21.01)

4. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to Time of Last Quantifiable Concentration (AUClast)
Description: AUClast of AZD0449 following intravenous administration of a single dose to healthy participants was assessed.
Time Frame: Part 1b: Day 1
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*nmol/L
Arm/Group | Part 1b (SAD IV) Cohort 1 | Part 1b (SAD IV) Cohort 2
Number analyzed (Participants) | 6 | 6
h*nmol/L | 3.567 (15.07) | 16.94 (20.39)

5. Primary Outcome: Area Under the Plasma Concentration Time Curve From Time Zero to 24 Hours After Dosing (AUC(0-24))
Description: AUC (0-24) of AZD0449 following intravenous administration of a single dose to healthy participants was assessed.
Time Frame: Part 1b: Day 1
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanomole/L (h*nmol/L)
Arm/Group | Part 1b (SAD IV) Cohort 1 | Part 1b (SAD IV) Cohort 2
Number analyzed (Participants) | 6 | 6
hour*nanomole/L (h*nmol/L) | 3.692 (14.31) | 17.03 (20.18)

6. Primary Outcome: Time to Reach Peak or Maximum Observed Concentration Following Drug Administration (Tmax)
Description: tmax of AZD0449 following intravenous administration of a single dose to healthy participants was assessed.
Time Frame: Part 1b: Day 1
Population: as for outcome 3
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 1b (SAD IV) Cohort 1 | Part 1b (SAD IV) Cohort 2
Number analyzed (Participants) | 6 | 6
Hours | 1.00 [0.73 to 1.00] | 0.69 [0.43 to 0.82]

7. Primary Outcome: Terminal Halflife, Estimated as (ln2)/-λz (t½λz )
Description: t½λz of AZD0449 following intravenous administration of a single dose to healthy participants was assessed.
Time Frame: Part 1b: Day 1
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Part 1b (SAD IV) Cohort 1 | Part 1b (SAD IV) Cohort 2
Number analyzed (Participants) | 6 | 6
Hours | 2.463 (0.5698) | 3.370 (2.453)

8. Primary Outcome: Total Body Clearance of Drug From Plasma After Intravascular Administration (CL)
Description: CL of AZD0449 following intravenous administration of a single dose of AZD0449 to healthy volunteers was assessed.
Time Frame: Part 1b: Day 1
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Liter/hour (L/h)
Arm/Group | Part 1b (SAD IV) Cohort 1 | Part 1b (SAD IV) Cohort 2
Number analyzed (Participants) | 6 | 6
Liter/hour (L/h) | 65.38 (9.099) | 57.05 (10.86)

9. Primary Outcome: Volume of Distribution for Parent Drug at Terminal Phase [Intravenous Administration] (λz)
Description: Vz of AZD0449 following intravenous administration of a single dose of AZD0449 to healthy volunteers was assessed.
Time Frame: Part 1b: Day 1
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | Part 1b (SAD IV) Cohort 1 | Part 1b (SAD IV) Cohort 2
Number analyzed (Participants) | 6 | 6
Liter | 232.0 (62.16) | 248.3 (109.0)

10. Primary Outcome: Terminal Rate Constant, Estimated by Loglinear Leastsquares Regression of the Terminal Part of the -Concentrationtime- Curve (λz)
Description: λz of AZD0449 following intravenous administration of a single dose to healthy participants was assessed.
Time Frame: Part 1b: Day 1
Population: as for outcome 3
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 1b (SAD IV) Cohort 1 | Part 1b (SAD IV) Cohort 2
Number analyzed (Participants) | 6 | 6
Hours | 0.285 [0.217 to 0.376] | 0.298 [0.084 to 0.371]

11. Primary Outcome: Time of Last Quantifiable Concentration (Tlast)
Description: tlast of AZD0449 following intravenous administration of a single dose to healthy participants was assessed.
Time Frame: Part 1b: Day 1
Population: as for outcome 3
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 1b (SAD IV) Cohort 1 | Part 1b (SAD IV) Cohort 2
Number analyzed (Participants) | 6 | 6
Hours | 9.98 [7.98 to 10.03] | 15.00 [11.98 to 24.03]

12. Primary Outcome: Dose Normalized Cmax (Cmax/D)
Description: Cmax/D of AZD0449 following intravenous administration of a single dose to healthy participants was assessed.
Time Frame: Part 1b: Day 1
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (nmol/L)/milligram (mg)
Arm/Group | Part 1b (SAD IV) Cohort 1 | Part 1b (SAD IV) Cohort 2
Number analyzed (Participants) | 6 | 6
(nmol/L)/milligram (mg) | 22.81 (15.95) | 28.65 (17.58)

13. Secondary Outcome: Number of Participants With Adverse Events and Serious Adverse Events
Description: Safety and tolerability of AZD0449 following intravenous administration of a single dose to healthy participants was assessed.
Time Frame: From screening up to follow-up visit [Part 1b (6±1 Days post-dose)]
Population: Safety Analysis Set included all participants who received at least one dose of AZD0449 and for whom any safety post-dose data were available.
Measure: Number; unit: Participants
Arm/Group | Part 1b (SAD IV) Cohort 1 | Part 1b (SAD IV) Cohort 2
Number analyzed (Participants) | 6 | 6
Participants
  Any Adverse Event (AE) | 2 | 2
  Any AE with outcome=death | 0 | 0
  Any serious AE (including events with outcome=death) | 0 | 0
  Any AE leading to withdrawal from study | 0 | 0
  Any AE leading to discontinuation of investigational medicinal product (IMP) | 0 | 0

14. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax)
Description: Cmax of AZD0449 following inhaled administration of single ascending doses of AZD0449, inhaled nebulized administration of multiple ascending doses to healthy participants and patients with mild asthma, and repeated inhaled administration to patients with mild asthma using a DPI was assessed.
Time Frame: Part 1a: Day 1, Part 2 and 3: Day 1 and Day 12
Population: The PK set consisted of all participants and patients who received at least one dose of AZD0449 and who had evaluable PK data, with no major protocol deviations thought to impact on the analysis of the PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomole/liter (nmol/L)
Arm/Group | Part 1a (SAD) Cohort 1 | Part 1a (SAD) Cohort 2 | Part 1a (SAD) Cohort 3 | Part 1a (SAD) Cohort 4 | Part 1a (SAD) Cohort 5 | Part 1a (SAD) Cohort 6 | Part 2a (MAD) Cohort 1 | Part 2a (MAD) Cohort 2 | Part 2b (MAD) Cohort 1 | Part 3a (DPI/PoM) | Part 3b (DPI/Healthy Participants)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 7 | 18 | 6
nanomole/liter (nmol/L)
  Day 1 | 0.4360 (54.69) | 1.791 (26.72) | 4.058 (68.59) | 8.646 (37.45) | 19.35 (20.56) | 26.13 (48.72) | 4.676 (18.64) | 12.09 (32.95) | 33.87 (39.92) | 12.34 (35.66) | 12.91 (29.36)
  Day 12 | NA (NA) — Cmax was not measured on Day 12 for Part 1. | NA (NA) — Cmax was not measured on Day 12 for Part 1. | NA (NA) — Cmax was not measured on Day 12 for Part 1. | NA (NA) — Cmax was not measured on Day 12 for Part 1. | NA (NA) — Cmax was not measured on Day 12 for Part 1. | NA (NA) — Cmax was not measured on Day 12 for Part 1. | 4.676 (39.84) | 13.12 (24.59) | 33.65 (39.61) | 16.32 (42.77) | 19.05 (39.71)

15. Secondary Outcome: Area Under the Plasma Concentration Time Curve From Time Zero to Infinity (AUCinf)
Description: AUCinf of AZD0449 following inhaled administration of single ascending doses of AZD0449, inhaled nebulized administration of multiple ascending doses to healthy participants and patients with mild asthma, and repeated inhaled administration to patients with mild asthma using a DPI was assessed.
Time Frame: Part 1a: Day 1, Part 2 and 3: Day 1 and Day 12
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*nmol/L
Arm/Group | Part 1a (SAD) Cohort 1 | Part 1a (SAD) Cohort 2 | Part 1a (SAD) Cohort 3 | Part 1a (SAD) Cohort 4 | Part 1a (SAD) Cohort 5 | Part 1a (SAD) Cohort 6 | Part 2a (MAD) Cohort 1 | Part 2a (MAD) Cohort 2 | Part 2b (MAD) Cohort 1 | Part 3a (DPI/PoM) | Part 3b (DPI/Healthy Participants)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 7 | 18 | 6
h*nmol/L
  Day 1 | 1.711 (58.87) | 4.964 (45.39) | 14.60 (127.6) | 35.61 (8.706) | 95.36 (33.47) | 141.2 (27.16) | 25.27 (16.74) | 57.82 (24.77) | 126.8 (48.59) | 82.44 (39.54) | 97.31 (30.03)
  Day 12: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6 | 7 | 18 | 6
  Day 12 |  |  |  |  |  |  | 84.73 (22.26) | 230.0 (22.39) | 615.8 (44.26) | 399.1 (46.09) | 658.9 (65.34)

16. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to Time of Last Quantifiable Concentration (AUClast)
Description: AUClast of AZD0449 following inhaled administration of single ascending doses of AZD0449, inhaled nebulized administration of multiple ascending doses to healthy participants and patients with mild asthma, and repeated inhaled administration to patients with mild asthma using a DPI was assessed.
Time Frame: Part 1a: Day 1, Part 2 and 3: Day 1 and Day 12
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*nmol/L
Arm/Group | Part 1a (SAD) Cohort 1 | Part 1a (SAD) Cohort 2 | Part 1a (SAD) Cohort 3 | Part 1a (SAD) Cohort 4 | Part 1a (SAD) Cohort 5 | Part 1a (SAD) Cohort 6 | Part 2a (MAD) Cohort 1 | Part 2a (MAD) Cohort 2 | Part 2b (MAD) Cohort 1 | Part 3a (DPI/PoM) | Part 3b (DPI/Healthy Participants)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 7 | 18 | 6
h*nmol/L
  Day 1 | 1.507 (64.24) | 4.608 (48.35) | 13.61 (127.2) | 32.17 (10.01) | 78.27 (28.58) | 121.8 (31.83) | 22.95 (13.65) | 52.67 (24.68) | 118.3 (49.99) | 74.54 (38.78) | 87.87 (31.91)
  Day 12: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6 | 7 | 18 | 6
  Day 12 |  |  |  |  |  |  | 61.90 (30.97) | 182.8 (29.08) | 509.6 (48.50) | 355.6 (48.27) | 570.5 (57.00)

17. Secondary Outcome: Area Under the Plasma Concentration Time Curve From Time Zero to 24 Hours After Dosing (AUC(0-24))
Description: AUC (0-24) of AZD0449 following inhaled administration of single ascending doses of AZD0449, inhaled nebulized administration of multiple ascending doses to healthy volunteers and patients with mild asthma, and repeated inhaled administration to patients with mild asthma using a DPI was assessed.
Time Frame: Part 1a: Day 1, Part 2 and 3: Day 1 and Day 12
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanomole/L (h*nmol/L)
Arm/Group | Part 1a (SAD) Cohort 1 | Part 1a (SAD) Cohort 2 | Part 1a (SAD) Cohort 3 | Part 1a (SAD) Cohort 4 | Part 1a (SAD) Cohort 5 | Part 1a (SAD) Cohort 6 | Part 2a (MAD) Cohort 1 | Part 2a (MAD) Cohort 2 | Part 2b (MAD) Cohort 1 | Part 3a (DPI/PoM) | Part 3b (DPI/Healthy Participants)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 7 | 18 | 6
hour*nanomole/L (h*nmol/L)
  Day 1 | 1.692 (58.94) | 4.798 (43.67) | 13.09 (118.0) | 29.46 (11.16) | 66.64 (27.05) | 94.029 (35.49) | 21.67 (13.03) | 50.07 (24.64) | 112.3 (50.33) | 69.00 (38.24) | 80.87 (31.67)
  Day 12: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6 | 7 | 18 | 6
  Day 12 |  |  |  |  |  |  | 27.39 (31.38) | 78.12 (32.39) | 166.4 (43.85) | 125.6 (48.14) | 167.9 (41.54)

18. Secondary Outcome: Time to Reach Peak or Maximum Observed Concentration Following Drug Administration (Tmax)
Description: tmax of AZD0449 following inhaled administration of single ascending doses of AZD0449, intravenous administration of a single dose to healthy volunteers, inhaled nebulized administration of multiple ascending doses to healthy volunteers and patients with mild asthma, and repeated inhaled administration to patients with mild asthma using a DPI was assessed.
Time Frame: Part 1a: Day 1, Part 2 and 3: Day 1 and Day 12
Population: as for outcome 3
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 1a (SAD) Cohort 1 | Part 1a (SAD) Cohort 2 | Part 1a (SAD) Cohort 3 | Part 1a (SAD) Cohort 4 | Part 1a (SAD) Cohort 5 | Part 1a (SAD) Cohort 6 | Part 2a (MAD) Cohort 1 | Part 2a (MAD) Cohort 2 | Part 2b (MAD) Cohort 1 | Part 3a (DPI/PoM) | Part 3b (DPI/Healthy Participants)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 7 | 18 | 6
Hours
  Day 1 | 1.00 [1.00 to 2.00] | 0.15 [0.13 to 0.37] | 0.10 [0.10 to 0.15] | 0.36 [0.22 to 1.50] | 0.34 [0.32 to 1.50] | 0.50 [0.33 to 2.02] | 0.20 [0.13 to 2.00] | 2.01 [0.23 to 2.13] | 0.43 [0.40 to 1.00] | 1.25 [0.23 to 3.02] | 2.00 [1.02 to 2.00]
  Day 12: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6 | 7 | 18 | 6
  Day 12 |  |  |  |  |  |  | 1.00 [0.12 to 2.00] | 0.23 [0.18 to 0.28] | 0.51 [0.37 to 2.00] | 1.58 [0.10 to 3.00] | 1.04 [1.00 to 3.00]

19. Secondary Outcome: Terminal Halflife, Estimated as (ln2)/-λz (t½λz )
Description: t½λz of AZD0449 following inhaled administration of single ascending doses of AZD0449, inhaled nebulized administration of multiple ascending doses to healthy volunteers and patients with mild asthma, and repeated inhaled administration to patients with mild asthma using a DPI was assessed.
Time Frame: Part 1a: Day 1, Part 2 and 3: Day 1 and Day 12
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Part 1a (SAD) Cohort 1 | Part 1a (SAD) Cohort 2 | Part 1a (SAD) Cohort 3 | Part 1a (SAD) Cohort 4 | Part 1a (SAD) Cohort 5 | Part 1a (SAD) Cohort 6 | Part 2a (MAD) Cohort 1 | Part 2a (MAD) Cohort 2 | Part 2b (MAD) Cohort 1 | Part 3a (DPI/PoM) | Part 3b (DPI/Healthy Participants)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 7 | 18 | 6
Hours
  Day 1 | 3.603 (1.281) | 6.049 (2.481) | 12.51 (5.169) | 24.07 (2.592) | 63.56 (30.66) | 84.26 (23.19) | 18.43 (6.029) | 18.35 (9.705) | 14.94 (3.707) | 14.93 (8.198) | 14.09 (2.7171)
  Day 12: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6 | 7 | 18 | 6
  Day 12 |  |  |  |  |  |  | 104.9 (43.78) | 115.2 (42.21) | 160.0 (63.96) | 124.4 (53.54) | 132.5 (33.23)

20. Secondary Outcome: Apparent Total Body Clearance of Drug From Plasma After Extravascular Administration (CL/F)
Description: CL/F of AZD0449 following inhaled administration of single ascending doses of AZD0449, inhaled nebulized administration of multiple ascending doses to healthy volunteers and patients with mild asthma, and repeated inhaled administration to patients with mild asthma using a DPI was assessed.
Time Frame: Part 1a: Day 1, Part 2 and 3: Day 1 and Day 12
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: liter/hour (L/h)
Arm/Group | Part 1a (SAD) Cohort 1 | Part 1a (SAD) Cohort 2 | Part 1a (SAD) Cohort 3 | Part 1a (SAD) Cohort 4 | Part 1a (SAD) Cohort 5 | Part 1a (SAD) Cohort 6 | Part 2a (MAD) Cohort 1 | Part 2a (MAD) Cohort 2 | Part 2b (MAD) Cohort 1 | Part 3a (DPI/PoM) | Part 3b (DPI/Healthy Participants)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 7 | 18 | 6
liter/hour (L/h)
  Day 1 | 168.5 (101.9) | 162.7 (73.35) | 259.2 (360.3) | 120.1 (10.39) | 93.84 (35.34) | 97.17 (26.31) | 128.0 (21.67) | 117.9 (26.32) | 113.0 (37.98) | 175.1 (87.78) | 141.9 (41.92)
  Day 12: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6 | 7 | 18 | 6
  Day 12 |  |  |  |  |  |  | 121.9 (44.38) | 88.89 (28.36) | 85.35 (29.74) | 118.4 (66.81) | 84.21 (28.88)

21. Secondary Outcome: Apparent Volume of Distribution for Parent Drug at Terminal Phase [Extravascular Administration] (Vz/F)
Description: Vz/F of AZD0449 following inhaled administration of single ascending doses of AZD0449, inhaled nebulized administration of multiple ascending doses to healthy volunteers and patients with mild asthma, and repeated inhaled administration to patients with mild asthma using a DPI was assessed.
Time Frame: Part 1a: Day 1, Part 2 and 3: Day 1 and Day 12
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | Part 1a (SAD) Cohort 1 | Part 1a (SAD) Cohort 2 | Part 1a (SAD) Cohort 3 | Part 1a (SAD) Cohort 4 | Part 1a (SAD) Cohort 5 | Part 1a (SAD) Cohort 6 | Part 2a (MAD) Cohort 1 | Part 2a (MAD) Cohort 2 | Part 2b (MAD) Cohort 1 | Part 3a (DPI/PoM) | Part 3b (DPI/Healthy Participants)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 7 | 18 | 6
Liter
  Day 1 | 818.1 (430.3) | 1275 (456.2) | 2696 (1301) | 4180 (620.1) | 8110 (3100) | 12080 (4962) | 3294 (779.9) | 3030 (1666) | 2542 (1340) | 3692 (2537) | 2977 (1280)
  Day 12: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6 | 7 | 18 | 6
  Day 12 |  |  |  |  |  |  | 20620 (18120) | 15970 (11290) | 20470 (13390) | 23520 (20930) | 15060 (3134)

22. Secondary Outcome: Terminal Rate Constant, Estimated by Loglinear Leastsquares Regression of the Terminal Part of the -Concentrationtime- Curve (λz)
Description: λz of AZD0449 following inhaled administration of single ascending doses of AZD0449, inhaled nebulized administration of multiple ascending doses to healthy volunteers and patients with mild asthma, and repeated inhaled administration to patients with mild asthma using a DPI was assessed.
Time Frame: Part 1a: Day 1, Part 2 and 3: Day 1 and Day 12
Population: as for outcome 14
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 1a (SAD) Cohort 1 | Part 1a (SAD) Cohort 2 | Part 1a (SAD) Cohort 3 | Part 1a (SAD) Cohort 4 | Part 1a (SAD) Cohort 5 | Part 1a (SAD) Cohort 6 | Part 2a (MAD) Cohort 1 | Part 2a (MAD) Cohort 2 | Part 2b (MAD) Cohort 1 | Part 3a (DPI/PoM) | Part 3b (DPI/Healthy Participants)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 7 | 18 | 6
Hours
  Day 1 | 0.210 [0.118 to 0.288] | 0.105 [0.079 to 0.243] | 0.055 [0.037 to 0.199] | 0.027 [0.026 to 0.035] | 0.013 [0.005 to 0.015] | 0.008 [0.005 to 0.012] | 0.041 [0.026 to 0.055] | 0.038 [0.021 to 0.113] | 0.053 [0.033 to 0.059] | 0.057 [0.017 to 0.084] | 0.048 [0.039 to 0.067]
  Day 12: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6 | 7 | 18 | 6
  Day 12 |  |  |  |  |  |  | 0.008 [0.003 to 0.009] | 0.006 [0.003 to 0.007] | 0.004 [0.002 to 0.006] | 0.005 [0.002 to 0.011] | 0.005 [0.003 to 0.007]

23. Secondary Outcome: Time of Last Quantifiable Concentration (Tlast)
Description: tlast of AZD0449 following inhaled administration of single ascending doses of AZD0449, inhaled nebulized administration of multiple ascending doses to healthy volunteers and patients with mild asthma, and repeated inhaled administration to patients with mild asthma using a DPI was assessed.
Time Frame: Part 1a: Day 1, Part 2 and 3: Day 1 and Day 12
Population: as for outcome 14
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 1a (SAD) Cohort 1 | Part 1a (SAD) Cohort 2 | Part 1a (SAD) Cohort 3 | Part 1a (SAD) Cohort 4 | Part 1a (SAD) Cohort 5 | Part 1a (SAD) Cohort 6 | Part 2a (MAD) Cohort 1 | Part 2a (MAD) Cohort 2 | Part 2b (MAD) Cohort 1 | Part 3a (DPI/PoM) | Part 3b (DPI/Healthy Participants)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 7 | 18 | 6
Hours
  Day 1 | 10.05 [6.00 to 11.98] | 17.99 [9.98 to 24.10] | 36.02 [9.98 to 36.13] | 48.19 [47.97 to 48.70] | 71.88 [71.58 to 72.05] | 144.41 [120.53 to 148.72] | 36.02 [35.95 to 36.10] | 36.00 [35.98 to 36.23] | 35.95 [35.92 to 35.98] | 36.02 [35.70 to 36.07] | 36.02 [36.00 to 36.05]
  Day 12: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6 | 7 | 18 | 6
  Day 12 |  |  |  |  |  |  | 168.03 [143.67 to 172.78] | 228.38 [167.73 to 242.13] | 359.96 [359.87 to 360.17] | 359.99 [263.87 to 360.45] | 360.00 [359.95 to 360.02]

24. Secondary Outcome: Dose Normalized Cmax (Cmax/D)
Description: Cmax/D of AZD0449 following inhaled administration of single ascending doses of AZD0449, inhaled nebulized administration of multiple ascending doses to healthy volunteers and patients with mild asthma, and repeated inhaled administration to patients with mild asthma using a DPI was assessed.
Time Frame: Part 1a: Day 1, Part 2 and 3: Day 1 and Day 12
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (nmol/L)/milligram (mg)
Arm/Group | Part 1a (SAD) Cohort 1 | Part 1a (SAD) Cohort 2 | Part 1a (SAD) Cohort 3 | Part 1a (SAD) Cohort 4 | Part 1a (SAD) Cohort 5 | Part 1a (SAD) Cohort 6 | Part 2a (MAD) Cohort 1 | Part 2a (MAD) Cohort 2 | Part 2b (MAD) Cohort 1 | Part 3a (DPI/PoM) | Part 3b (DPI/Healthy Participants)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 7 | 18 | 6
(nmol/L)/milligram (mg)
  Day 1 | 4.589 (54.69) | 6.396 (26.72) | 4.831 (68.59) | 5.404 (37.45) | 6.047 (20.56) | 5.226 (48.72) | 3.897 (18.64) | 4.837 (32.95) | 6.775 (39.92) | 2.468 (35.66) | 2.582 (29.36)
  Day 12: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6 | 7 | 18 | 6
  Day 12 |  |  |  |  |  |  | 3.897 (39.84) | 5.248 (24.59) | 6.730 (39.61) | 3.265 (42.77) | 3.811 (39.71)

25. Secondary Outcome: Change From Baseline in 2 Hours Post-dose Fractional Excretion of Nitric Oxide (FeNO)
Description: Assessment of anti-inflammatory effect by evaluating change from baseline in FeNO, 2 hours post-dose of AZD0449 in patients with mild asthma was assessed.
Time Frame: At Baseline and Day 12
Population: The Full Analysis Set (FAS) consisted of all participants randomized into the study who have received at least 1 dose of IMP and having at least one 2-hour post-dose FeNO assessment after the first IMP intake.
Measure: Least Squares Mean (90% Confidence Interval); unit: parts per billion (ppb)
Arm/Group | Part 2a (MAD) Cohort 1 | Part 2a (MAD) Cohort 2 | Part 2a (MAD) Placebo | Part 3a (DPI/PoM) | Part 3a (DPI/PoM) Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 18 | 18
parts per billion (ppb) | -22.6 [-31.4 to -13.8] | -22.2 [-30.9 to -5.49] | -14.3 [-23.1 to -5.49] | -15.0 [-18.9 to -11.1] | -12.0 [-15.9 to -8.03]
Statistical Analysis 1: Comparison: Part 2a (MAD) Cohort 1 vs Part 2a (MAD) Cohort 2; Comparison of Part 2a (MAD) Cohort 1 Vs Part 2a (MAD) Cohort 2; Test type: Other; p = 0.9511, Linear Mixed Model; LS means difference = -0.440, 90% CI 2-sided [-12.9 to 12.0]
Statistical Analysis 2: Comparison: Part 2a (MAD) Cohort 2 vs Part 2a (MAD) Placebo; Comparison of Part 2a (MAD) Cohort 2 Vs Part 2a (MAD) Placebo; Test type: Other; p = 0.2849, Linear Mixed Model; LS means difference = -7.87, 90% CI 2-sided [-20.3 to 4.59]
Statistical Analysis 3: Comparison: Part 2a (MAD) Cohort 1 vs Part 2a (MAD) Placebo; Comparison of Part 2a (MAD) Cohort 1 Vs Part 2a (MAD) Placebo; Test type: Other; p = 0.2595, Linear Mixed Model; LS means difference = -8.31, 90% CI 2-sided [-20.8 to 4.14]
Statistical Analysis 4: Comparison: Part 3a (DPI/PoM) vs Part 3a (DPI/PoM) Placebo; Comparison of Part 3a (DPI/PoM) Vs Part 3a (DPI/PoM) Placebo; Test type: Other; p = 0.3604, Linear Mixed Model; LS means difference = -3.04, 90% CI 2-sided [-8.60 to 2.51]

26. Secondary Outcome: Change From Baseline in 2 Hours Post-dose in FeNO (AUC (0-12))
Description: Assessment of anti-inflammatory effect by evaluating change from baseline in FeNO (AUC (0-12)), 2 hours post-dose of AZD0449 in patients with mild asthma was assessed.
Time Frame: At Baseline and Day 12
Population: as for outcome 25
Measure: Least Squares Mean (90% Confidence Interval); unit: parts per billion (ppb)
Arm/Group | Part 2a (MAD) Cohort 1 | Part 2a (MAD) Cohort 2 | Part 2a (MAD) Placebo | Part 3a (DPI/PoM) | Part 3a (DPI/PoM) Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 18 | 18
parts per billion (ppb) | -299 [-399 to -200] | -274 [-373 to -174] | -200 [-300 to -101] | -213 [-250 to -176] | -162 [-199 to -126]
Statistical Analysis 1: Comparison: Part 2a (MAD) Cohort 1 vs Part 2a (MAD) Cohort 2; Comparison of Part 2a (MAD) Cohort 1 Vs Part 2a (MAD) Cohort 2; Test type: Other; p = 0.7544, Linear Mixed Model; LS means difference = -25.4, 90% CI 2-sided [-166 to 115]
Statistical Analysis 2: Comparison: Part 2a (MAD) Cohort 2 vs Part 2a (MAD) Placebo; Comparison of Part 2a (MAD) Cohort 2 Vs Part 2a (MAD) Placebo; Test type: Other; p = 0.3750, Linear Mixed Model; LS means difference = -73.3, 90% CI 2-sided [-214 to 67.6]
Statistical Analysis 3: Comparison: Part 2a (MAD) Cohort 1 vs Part 2a (MAD) Placebo; Comparison of Part 2a (MAD) Cohort 1 Vs Part 2a (MAD) Placebo; Test type: Other; p = 0.2377, Linear Mixed Model; LS means difference = -98.7, 90% CI 2-sided [-240 to 42.3]
Statistical Analysis 4: Comparison: Part 3a (DPI/PoM) vs Part 3a (DPI/PoM) Placebo; Comparison of Part 3a (DPI/PoM) Vs Part 3a (DPI/PoM) Placebo; Test type: Other; p = 0.1105, Linear Mixed Model; LS means difference = -50.4, 90% CI 2-sided [-102 to 1.61]

ADVERSE EVENTS:
Time Frame: From screening up to follow-up visit [Part 1 a/b (6±1 Days post-dose)] [Part 2a (Day 22±1 (10±1 days post-last dose)], Safety Monitoring Period 2b/3a [Day 17 to 27 (15 day post-last dose)].
Arm/Group | Part 1a (SAD) Placebo | Part 1a (SAD) Cohort 1 | Part 1a (SAD) Cohort 2 | Part 1a (SAD) Cohort 3 | Part 1a (SAD) Cohort 4 | Part 1a (SAD) Cohort 5 | Part 1a (SAD) Cohort 6 | Part 1b (SAD IV) Cohort 1 | Part 1b (SAD IV) Cohort 2 | Part 2a (MAD) Placebo | Part 2a (MAD) Cohort 1 | Part 2a (MAD) Cohort 2 | Part 2b (MAD) Placebo | Part 2b (MAD) Cohort 1 | Part 3a (DPI/PoM) Placebo | Part 3a (DPI/PoM) | Part 3b (DPI/Healthy Participants) Placebo | Part 3b (DPI/Healthy Participants)
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/2 | 0/7 | 0/18 | 0/18 | 0/2 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/2 | 0/7 | 0/18 | 0/18 | 0/2 | 0/6
Other Adverse Events (participants affected / at risk) | 3/12 | 2/6 | 2/6 | 3/6 | 3/6 | 3/6 | 1/6 | 2/6 | 2/6 | 4/6 | 5/6 | 3/6 | 2/2 | 6/7 | 15/18 | 14/18 | 0/2 | 3/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1a (SAD) Placebo (N=12) | Part 1a (SAD) Cohort 1 (N=6) | Part 1a (SAD) Cohort 2 (N=6) | Part 1a (SAD) Cohort 3 (N=6) | Part 1a (SAD) Cohort 4 (N=6) | Part 1a (SAD) Cohort 5 (N=6) | Part 1a (SAD) Cohort 6 (N=6) | Part 1b (SAD IV) Cohort 1 (N=6) | Part 1b (SAD IV) Cohort 2 (N=6) | Part 2a (MAD) Placebo (N=6) | Part 2a (MAD) Cohort 1 (N=6) | Part 2a (MAD) Cohort 2 (N=6) | Part 2b (MAD) Placebo (N=2) | Part 2b (MAD) Cohort 1 (N=7) | Part 3a (DPI/PoM) Placebo (N=18) | Part 3a (DPI/PoM) (N=18) | Part 3b (DPI/Healthy Participants) Placebo (N=2) | Part 3b (DPI/Healthy Participants) (N=6)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 1 (1) | 2 (4) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (4) | 2 (6) | 1 (2) | 1 (3) | 3 (5) | 6 (10) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (7) | 2 (3) | 1 (1) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (5) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear discomfort (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SARS-CoV-2 antibody test positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 | 0 (0) | 0 (0) | 0 (0)
Abnormal dreams (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (5) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness postural (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eructation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 2 (3) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Facial pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hordeolum (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Forced expiratory volume decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aphthous ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram T wave abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Burning sensation mucosal (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Taste disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Testis discomfort (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catarrh (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Application site rash (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 1 (1)
Application site dermatitis (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Application site irritation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Catheter site rash (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infusion site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infusion site rash (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Skin fissures (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Macule (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Nasal injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Animal scratch (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lip injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Allergy to arthropod bite (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Depressed mood (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
External ear inflammation (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Photopsia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No unpublished information may be disclosed without prior written approval from AstraZeneca AB.

DOCUMENTS (2):
  • Study Protocol (2021-02-04): https://cdn.clinicaltrials.gov/large-docs/99/NCT03766399/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-05): https://cdn.clinicaltrials.gov/large-docs/99/NCT03766399/SAP_001.pdf